CLINICAL TRIAL: NCT03413384
Title: A Randomized, Double Blinded, Placebo-controlled Phase II Study to Assess the Efficacy and Safety of Ceftriaxone in Patients With Mild to Moderate Parkinson's Disease Dementia
Brief Title: To Assess the Efficacy and Safety of Ceftriaxone in Patients With Mild to Moderate Parkinson's Disease Dementia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BrainX Corporation (Industry)
Collaborators: Virginia Contract Research Organization Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRICEFA20170414
Record Dates: First submitted 2018-01-08; First posted 2018-01-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease Dementia
Keywords: Parkinson's Disease; Parkinson's Disease Dementia
MeSH Terms: conditions — Parkinson Disease | interventions — Ceftriaxone; Injections, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ceftriaxone (Experimental): 1. Name: Ceftriaxone
  2. Dosage form: crystalline powder for intramuscular injection
  3. Dose(s): 1 g
  4. Dosing schedule: 1 g ceftriaxone with around 2.0 ml of lidocaine solvent per day for Day 1, 3, and 5 per cycle on a 2 weekly cycle
  Interventions: Drug: Ceftriaxone
- Placebo (Placebo Comparator): same amount volume of placebo will be given on Day 1, Day 3, and Day 5 per cycle on a 2 weekly cycle
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ceftriaxone — 1 g ceftriaxone per day for Day 1, 3, and 5 per cycle on a 2 weekly cycle
  Other Names: Ceftriaxone Sandoz powder for IV Injection
  Arms: Ceftriaxone
Other: Placebo — Placebo per day for Day 1, 3, and 5 per cycle on a 2 weekly cycle
  Arms: Placebo

SUMMARY:
This is a randomized, double blinded, placebo-controlled Phase II study to investigate the efficacy and safety of ceftriaxone in patients with mild to moderate Parkinson's disease dementia (PDD).This study will enroll approximately 106 patients to have up to 84 evaluable subjects, and conduct in Chung Shan Medical University Hospital, National Taiwan University Hospital, Kaohsiung Chang Gung Memorial Hospital, China Medical University Hospital, Changhua Christian Hospital, and Taipei Veterans General Hospital.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disorder that can cause significant disability and decrease quality of life. It is a chronic and progressive disease which means the symptoms become worse over time.

Parkinson's disease dementia (PDD) is a decline in thinking and reasoning that develops in many people living with PD at least a year after diagnosis. An estimated 50 to 80 percent of patients with PD eventually experience dementia as the disease progresses. Ceftriaxone is a kind of antibiotics, which has been marketed in many countries. This is the first time for ceftraxone treatment on PDD patient. The primary objective of this Phase II study is to evaluate the improvement of cognitive function in PDD patients with ceftriaxone administration.

This study will enroll approximately 106 patients, and conduct in multiple hospitals in Taiwan. Recruitment number of each site will be adjusted according to its enrollment status under the competitive enrollment model. Subjects will receive either ceftriaxone or placebo in a 1:1 ratio. One of the subjects' main caregiver should be involved to get the information of function of daily life and help to complete scale evaluation.

The study lasts about 33 weeks, during which eligible patients will be given 1 g/day/dose of ceftriaxone or placebo via injection 3 doses every cycle (2 weekly cycle), for a total of 16 cycles. And the subjects can choose to get injection either in the clinical site or in their house.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are male or female, age 50-85 years, inclusive.
2. Diagnosis of idiopathic Parkinson's disease (PD) based on the UK Parkinson's Disease Society Brain Bank Criteria and with a modified Hoehn and Yahr Stage of I to IV.
3. Patients have been receiving stable dose of medications equivalent up to 1800 mg/day of levodopa for Parkinson's disease at least 2 weeks prior to screening and patients are considered as being optimally treated at screening and no known further adjustments of current medication needed to improve the subject's status of PD during the study period by the judgment of the Investigator based on the subject's history, previous treatments, and the clinical presentation.
4. Diagnosis of PDD based on Movement Disorder Society (MDS) Task Force criteria as the following items:

   1. A diagnosis of PD based on UK Parkinson's Disease Society Brain Bank Criteria
   2. PD development prior to the onset of dementia based on patient/caregiver history or records
   3. Cognitive deficiency severe enough to impair daily life based on patient/caregiver interview or questionnaire
   4. Impairment of at least 2 of the following domains: attention, executive function, visuo-constructive ability, memory Besides, patients' Mini-Mental State Examination (MMSE) should be in the range of 18-25 (inclusive) or CDR scale in the range of 0.5-2. Note that MMSE range 16-25 for illiterate. Illiterate is defined as no education history.
5. Patients who are eligible and able to participate in the study must be judged by the investigator to evaluate the competency of providing informed consent for this dementia related study (the decision making is based on MacArthur Competence Assessment concept) and should be able to understand the language in which the tests require so and must be able to perform all the assessments.
6. All male and female patients with child-bearing potential (between puberty and 2 years after menopause) should use at least any one of the appropriate contraception methods shown below, for during and at least 4 weeks after ceftriaxone treatment.

   1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception).
   2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   3. Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
   4. Combination of any two of the following listed methods: (d.1+d.2 or d.1+d.3, or d.2+d.3):

   d.1 Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

   d.2 Placement of an intrauterine device (IUD) or intrauterine system (IUS). d.3 Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Exclusion Criteria:

1. Any indication of forms of Parkinsonism other than idiopathic PD.
2. Diagnosis of possible PDD.
3. Diagnosis of dementia with Lewy Bodies.
4. Mental/physical/social condition which could preclude performing efficacy or safety assessments.
5. Medical history of brain or other clinically significant neurological/psychiatric disorders or injuries other than PD or PDD that would hinder or interfere the study safety or efficacy evaluation in the opinion of the Investigator.
6. The patients have received neurosurgical intervention related to PD (e.g. deep brain stimulation (DBS), thalamotomy etc.) or are scheduled to do so during the trial period.
7. The patients have history of allergic response to levodopa, ceftriaxone, cephalosporin class of drugs or ursodiol or lidocaine.
8. Malignant neoplastic disease, either currently active or in remission for less than 1 year.
9. Clinically significant and unstable gastrointestinal, renal, endocrine, pulmonary, or cardiovascular disease, including not well controlled hypertension, asthma, chronic obstructive pulmonary disease, diabetes, hyperbilirubinemia, impaired vitamin K synthesis or low vitamin K stores that would hinder or interfere participation to the study in the opinion of the Investigator.
10. Patients with abdominal ultrasound examination imaging shows active biliary obstruction disease at PI's discretion during screening.
11. The patients are currently experiencing unpredictable or intractable or troublesome dyskinesia or fluctuations in their symptoms.
12. Patients with the following medications that could put patients at risk, interfere with study evaluations, or prevent meeting the requirements of the study at the judgement of PI should be excluded :

    1. Centrally acting anticholinergic medication currently or within 4 weeks prior to the screening visit.
    2. Cocaine, opioids, ethanol (binge drinking or heavy alcohol defined by SAMHSA and NIAAA) currently or within 4 weeks prior to the screening visit; amphetamines, cannabinoids abuse history or taking currently or within 3 months prior to the screening visit.
    3. Acetylcholinesterase inhibitors or memantine currently or within 4 weeks prior to the screening visit, except that patients have been stable controlled and have been receiving stable dose of the acetylcholinesterase inhibitors or memantine for at least 4 weeks prior to screening or are considered being optimally treated at screening without further dose adjustments needed as judged by the Investigator.
    4. Ceftriaxone or cephalosporin or penicillin or β-lactam currently or within 4 weeks prior to the screening visit.
    5. Neuroleptics or antipsychotics for treatment of psychotic symptoms (e.g., hallucinations) within 4 weeks prior to the screening visit, except that patients have been stable controlled and have been receiving stable dose of the neuroleptics or antipsychotics for at least 4 weeks prior to screening or are considered being optimally treated at screening without further dose adjustments needed as judged by the Investigator.
    6. A drug that has severe hepatotoxic or renal toxic within 4 weeks prior to the screening visit.
    7. Warfarin, cyclosporin, vancomycin, amsacrine, aminoglycosides, fluconazole, chloramphenicol currently or within 4 weeks prior to the screening visit.
13. Currently participating in another clinical trial or who participated in a previous clinical trial and received any investigational product treatment within 4 weeks prior to the screening visit.
14. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer from such.
15. Patients who are not able to take MRI and TRODAT SPECT examination.
16. Patients who are pregnant or breast feeding.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare the treatment difference in mean net change in ADAS-Cog score with time course | from baseline to week 17 and 33 visits
  ADAS-Cog is a validated instrument to assess dementia covering memory, orientation, language, praxis and consisting of 11 items. The total possible scores range from 70 (severe impairment) to 0 (no impairment).

SECONDARY OUTCOMES:
Changes in Unified Parkinson's Disease Rating Scale (UPDRS) score | from baseline to week 17 and 33 visits
  The UPDRS system is a composite scale intended for rating patients with PD. Scores are rated as 0-4 (0-1 for some Part IV), representing 0=normal and 1 or 4=maximal deficit, symptoms, or impairment.
Changes in Judgment of Line Orientation score | from baseline to week 17 and 33 visits
  The Judgment of Line Orientation (JLO) test is a widely used measure of visuospatial judgment. A score of 17 or less is considered a sign of severe deficit.
Changes in Mini-Mental State Examination (MMSE) score | from baseline at week 17 and 33 visits
  The MMSE is a brief, quantitative measure of cognitive status in adults. The instrument examines orientation, registration, attention, calculation, recall, visuo-spatial abilities and language. The maximum score is 30, with higher scores indicating better cognitive function.
Changes in Clinical Dementia Rating (CDR) Scale score | from baseline to week 17 and 33 visits
  The CDR Scale is a 5-point scale used to characterize 6 domains of cognitive and functional performance applicable to related dementias: memory, orientation, judgment & problem solving, community affairs, home & hobbies, and personal care. This score is useful for characterizing and tracking a patient's level of impairment/dementia with 0=normal, 0.5 =very mild dementia, 1=mild dementia, 2=moderate dementia, 3=severe dementia.
Changes in Color Trail Test score | from baseline to week 17 and 33 visits
  Color Trail Test provides quantitative and qualitative information by two trials. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors.
Changes in MRI image for atrophy rate of brain | from baseline to week 17 and 33 visits
  Multimodal MRI examinations will be performed on a 3T MRI scanner with a standard 8-channel head coil. Region of interest in the brain will be evaluated for functional changes including atrophy rate from baseline data.
Changes in MRI image for dopaminergic projection from substantia nigra to striatum | from baseline to week 17 and 33 visits
  Multimodal MRI examinations will be performed on a 3T MRI scanner with a standard 8-channel head coil. Region of interest in the brain will be evaluated for functional changes including dopaminergic projection from baseline data.
Changes in Tc-99m TRODAT SPECT image | from baseline to week 17 and 33 visits
  SPECT assessment will use Tc-99m, a radio tracer with high selectivity and specificity for the striatum dopamine transporter (DAT) density evaluation. DAT density change from baseline will be calculated from region of interest drawn in the striatum by independent readers.

OTHER OUTCOMES:
Net change of biomarker α-synuclein data | from baseline to week 17 and 33 visits
  Patients' plasma samples will be collected to analyze α-synuclen by immunomagnetic reduction (IMR) assay kit developed by Magqu Company.
Net change of biomarker Aβ42 data | from baseline to week 17 and 33 visits
  Patients' plasma samples will be collected to analyze α-synuclen by immunomagnetic reduction (IMR) assay kit developed by Magqu Company.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Ho, Study Director — China Medical University, China
Locations (6):
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Kaohsiung
  - Chung Shan Medical University Hospital, Taichung, Taichung
  - China Medical University Hospital, Taichung, Taichung
  - National Taiwan University Hospital, Taipei, Taipei
  - Taipei Veterans General Hospital, Taipei, Taipei
  - Changhua Christian Hospital, Changhua

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arlet J. [40 years of the "Revue du Rhumatisme" (1947-1987). Contribution of French rheumatologists to progress in rheumatology]. Rev Rhum Mal Osteoartic. 1989 Apr;56(5):355-67. No abstract available. French. PMID 2658001